CLINICAL TRIAL: NCT01883063
Title: PATIENT OUTCOME COMPARISON OF INTRAMEDULLARY LOCKED NAILING VERSUS NONOPERATIVE MANAGEMENT OF EXTRA-ARTICULAR AND MINIMALLY DISPLACED INTRA-ARTICULAR DISTAL RADIUS FRACTURES IN THE ELDERLY
Brief Title: Distal Radius Fracture - Treatment Comparison
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Enrollment
Sponsor: Sonoma Orthopedic Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRx-001
Record Dates: First submitted 2013-06-14; First posted 2013-06-21 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Minimally Displaced Intra-articular Distal Radius Fracture
MeSH Terms: interventions — Surgical Procedures, Operative; Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WRx™ Intramedullary Nail (Experimental): Patients in this arm of the study will be treated with a minimally invasive WRx™ Intramedullary Nail for their wrist fracture.
  Interventions: Device: Surgical Treatment
- Non surgical treatment (Cast) (Active Comparator): Patients in this arm of the study will be treated with a cast for their wrist fracture.
  Interventions: Device: Non surgical Treatment (Cast or splint)

INTERVENTIONS:
Device: Surgical Treatment — Patients will be treated for distal radius fractures surgically with a WRx™ Intramedullary Nail
  Arms: WRx™ Intramedullary Nail
Device: Non surgical Treatment (Cast or splint) — Patients will be treated for distal radius fractures non surgically with a cast or splint
  Arms: Non surgical treatment (Cast)

SUMMARY:
This is a prospective multi-site study. Subjects with distal radius fractures will be enrolled. Subjects will be treated surgically with a Sonoma WRx™ device or managed non-operatively with a splint or cast. Subjects will be enrolled in each group according to physician's standard of care (either casting/splinting or surgery) for distal radius fractures. Subjects will be enrolled based on the study's inclusion/exclusion criteria with a final qualifying decision made by a group of three independent adjudicators. The final qualifying review should allow for similar patient groups within each arm of the study due to the variability that can arise in fracture classification. Review by the adjudicators should be completed within 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Closed extra-articular distal radius fracture or a minimally displaced intra-articular fracture
* Fracture classified as an AO/OTA A2, A3, C1 or C2 with or without an ulnar styloid fracture
* Must be treated within the first 14 days of injury,
* Male or female greater than or equal to 65 years of age.
* Able to understand the requirements of the study, provide a written informed consent and comply with the study protocol
* Ability to understand and provide written authorization for use and disclosure of personal health information
* Fracture that can be treated closed with or without closed reduction

Exclusion Criteria:

* Concomitant contralateral or ipsilateral upper extremity fractures
* Ipsilateral ulna (excluding styloid) fracture
* Open fracture
* Previous ipsilateral distal radius fracture in the 2 years prior to enrollment with deformity
* Unstable distal radioulnar joint after fracture fixation
* Fractures where the transverse fracture line is less than 10mm from the distal radius joint surface
* Artery or Nerve injury secondary to fracture
* History of alcoholism
* Currently on chemotherapy or radiation therapy
* Currently on worker's compensation
* Rheumatoid arthritis or other inflammatory arthropathies.
* History of chronic pain issues or psychiatric disorder that precludes reliable follow-up.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Composite Patient Outcomes Over Time | Data will be collected at 2, 6, 12, 26, 52 weeks
  Patient outcomes will be measured with the DASH, PRWE and a patient questionnaire.

SECONDARY OUTCOMES:
Change in Composite Functional Outcomes Over Time | Data will be collected at 2, 6, 12, 26, 52 weeks
  Measurements of range of motion, strength and fracture healing will be used to determine functional outcomes.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Cadence Health, Winfield, Illinois
  - University of Missouri, Columbia, Missouri
  - John Peter Smith Hospital, Fort Worth, Texas